CLINICAL TRIAL: NCT02488005
Title: The Use of Small Bowel Ultrasound to Predict Response to Remicade Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 15-0878
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
Keywords: Inflammatory Bowel Disease; Small Bowel; Crohn's Disease; Small Bowel Ultrasound
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Small Bowel Ultrasound (Experimental): Subjects will receive a small bowel ultrasound to measure bowel wall thickness at Week 0 and Week 14
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — An ultrasound of the small bowel will be done by a radiologist or ultrasound technician. Subject should not eat or drink anything (i.e. no food and no water/beverages) for 8 hours prior to their ultrasound appointment

SUMMARY:
Small bowel ultrasound (SBUS) is emerging as a well tolerated, non-invasive, radiation free, low cost measure to assess inflammatory bowel disease (IBD), and is being used as first-line imaging in Europe. SBUS findings have been shown to correlate with endoscopic findings, and a small number of recent studies have looked at change in bowel wall thickness (BWT) in response to anti-tumor necrosis factor (anti-TNF) therapy. However, the use of SBUS to detect response to anti-TNF therapy has not been tested in pediatric patients. The purpose of this study is to apply the use of SBUS to pediatric patients with Crohn's disease and to assess response to treatment with infliximab. The investigators will also measure C-reactive protein and fecal calprotectin at baseline, and additionally measuring IFX levels and anti-infliximab antibodies (ATI) at week 14 to assess change in biochemical response to infliximab treatment, as well as correlation between these markers with changes in patient reported outcomes via a weighted pediatric Crohn's disease activity questionnaire (wPCDAI) and changes in BWT. This study is novel in that it will be the first study in pediatric patients to use SBUS to assess response to IFX therapy, and will also be the first study to correlate SBUS findings with therapeutic drug monitoring (TDM). This study has the potential to propagate the use of SBUS in the pediatric population, as the use of TDM in concert with small bowel imaging post-induction will allow the investigators to tailor therapy early in the treatment course.

DETAILED DESCRIPTION:
Pediatric inflammatory bowel disease (IBD) patients are at increased risk for high ionizing radiation exposure in the assessment of their condition. Small bowel ultrasound (SBUS) is emerging as a well tolerated, non-invasive, radiation free, low cost measure to assess inflammatory bowel disease, and is being used as first-line imaging in Europe. SBUS findings have been shown to correlate with endoscopic findings, and a small number of recent studies have looked at change in bowel wall thickness (BWT), in response to anti-TNF therapy.

The use of SBUS to detect response to anti-TNF therapy has not been tested in pediatric patients. In addition, these studies frequently use Crohn's Disease Activity Index (CDAI) as a measure of clinical activity, yet it is known from multiple studies including the SONIC trial that CDAI is not a reliable or accurate measure to predict mucosal healing. A weighted PCDAI will be used instead, which has been shown to perform better than the original PCDAI and is more feasible, especially considering the study spans 14 weeks and scoring items such as height velocity from the full PCDAI will be irrelevant.

The goal of this study is to measure bowel wall thickness (BWT) prior to initiating infliximab (IFX 0) and at week 14 and to look at the correlation between change in BWT (delta BWT) with change in clinical disease activity (delta wPCDAI) between these two time points. The research team will measure fecal calprotectin at baseline and at week 14 with stool collected the day prior to the visit using a specimen collection kit given to subjects. The research team will also collect results from routine laboratories (including C-Reactive Protein, Erythrocyte Sedimentation Rate, Complete Blood Count, and Albumin) done before each infusion, and IFX levels and anti-infliximab antibodies (ATI) at week 14 to assess change in biochemical response to infliximab treatment, as well as correlation between these markers with changes in patient reported outcomes (via a wPCDAI questionnaire) and changes in BWT.

ELIGIBILITY:
Inclusion Criteria:

* No infliximab therapy previously initiated
* Infliximab indicated for treatment of IBD
* Patient consent/assent and/or parent/guardian consent
* Ability to remain in follow-up for 14 weeks from start of study

Exclusion Criteria:

* Lack of small bowel disease
* Inability to give consent or adhere to study protocol
* Infliximab-experienced
* Presence of active infections
* Presence of abscess or strictures
* Current or planned Pregnancy for the 14 week study duration

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla C. Dubinsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Susan and Leonard Feinstein Inflammatory Bowel Disease Clinical Center, New York, New York, United States

REFERENCES:
- [Background] Sauer CG, Kugathasan S, Martin DR, Applegate KE. Medical radiation exposure in children with inflammatory bowel disease estimates high cumulative doses. Inflamm Bowel Dis. 2011 Nov;17(11):2326-32. doi: 10.1002/ibd.21626. Epub 2011 Jan 13. PMID 21987300
- [Background] Panes J, Bouhnik Y, Reinisch W, Stoker J, Taylor SA, Baumgart DC, Danese S, Halligan S, Marincek B, Matos C, Peyrin-Biroulet L, Rimola J, Rogler G, van Assche G, Ardizzone S, Ba-Ssalamah A, Bali MA, Bellini D, Biancone L, Castiglione F, Ehehalt R, Grassi R, Kucharzik T, Maccioni F, Maconi G, Magro F, Martin-Comin J, Morana G, Pendse D, Sebastian S, Signore A, Tolan D, Tielbeek JA, Weishaupt D, Wiarda B, Laghi A. Imaging techniques for assessment of inflammatory bowel disease: joint ECCO and ESGAR evidence-based consensus guidelines. J Crohns Colitis. 2013 Aug;7(7):556-85. doi: 10.1016/j.crohns.2013.02.020. Epub 2013 Apr 11. PMID 23583097
- [Background] Calabrese E, Zorzi F, Zuzzi S, Ooka S, Onali S, Petruzziello C, Lasinio GJ, Biancone L, Rossi C, Pallone F. Development of a numerical index quantitating small bowel damage as detected by ultrasonography in Crohn's disease. J Crohns Colitis. 2012 Sep;6(8):852-60. doi: 10.1016/j.crohns.2012.01.015. Epub 2012 Feb 23. PMID 22398077
- [Background] Onali S, Calabrese E, Petruzziello C, Zorzi F, Sica GS, Lolli E, Ascolani M, Condino G, Pallone F, Biancone L. Endoscopic vs ultrasonographic findings related to Crohn's disease recurrence: a prospective longitudinal study at 3 years. J Crohns Colitis. 2010 Sep;4(3):319-28. doi: 10.1016/j.crohns.2009.12.010. Epub 2010 Feb 19. PMID 21122521
- [Background] Zorzi F, Stasi E, Bevivino G, Scarozza P, Biancone L, Zuzzi S, Rossi C, Pallone F, Calabrese E. A sonographic lesion index for Crohn's disease helps monitor changes in transmural bowel damage during therapy. Clin Gastroenterol Hepatol. 2014 Dec;12(12):2071-7. doi: 10.1016/j.cgh.2014.04.036. Epub 2014 May 6. PMID 24813174
- [Background] Castiglione F, Testa A, Rea M, De Palma GD, Diaferia M, Musto D, Sasso F, Caporaso N, Rispo A. Transmural healing evaluated by bowel sonography in patients with Crohn's disease on maintenance treatment with biologics. Inflamm Bowel Dis. 2013 Aug;19(9):1928-34. doi: 10.1097/MIB.0b013e31829053ce. PMID 23835441
- [Background] Moreno N, Ripolles T, Paredes JM, Ortiz I, Martinez MJ, Lopez A, Delgado F, Moreno-Osset E. Usefulness of abdominal ultrasonography in the analysis of endoscopic activity in patients with Crohn's disease: changes following treatment with immunomodulators and/or anti-TNF antibodies. J Crohns Colitis. 2014 Sep;8(9):1079-87. doi: 10.1016/j.crohns.2014.02.008. Epub 2014 Mar 7. PMID 24613399
- [Background] Paredes JM, Ripolles T, Cortes X, Martinez MJ, Barrachina M, Gomez F, Moreno-Osset E. Abdominal sonographic changes after antibody to tumor necrosis factor (anti-TNF) alpha therapy in Crohn's Disease. Dig Dis Sci. 2010 Feb;55(2):404-10. doi: 10.1007/s10620-009-0759-7. Epub 2009 Mar 7. PMID 19267199
- [Background] Turner D, Griffiths AM, Walters TD, Seah T, Markowitz J, Pfefferkorn M, Keljo D, Waxman J, Otley A, LeLeiko NS, Mack D, Hyams J, Levine A. Mathematical weighting of the pediatric Crohn's disease activity index (PCDAI) and comparison with its other short versions. Inflamm Bowel Dis. 2012 Jan;18(1):55-62. doi: 10.1002/ibd.21649. Epub 2011 Feb 23. PMID 21351206
- [Derived] Dolinger MT, Choi JJ, Phan BL, Rosenberg HK, Rowland J, Dubinsky MC. Use of Small Bowel Ultrasound to Predict Response to Infliximab Induction in Pediatric Crohn's Disease. J Clin Gastroenterol. 2021 May-Jun 01;55(5):429-432. doi: 10.1097/MCG.0000000000001367. PMID 32453126

RESULTS

PARTICIPANT FLOW:
Groups:
- Small Bowel Ultrasound: Subjects had a small bowel ultrasound done by a radiologist or ultrasound technician to measure bowel wall thickness at Week 0 and Week 14.
Period: Overall Study
Arm/Group | Small Bowel Ultrasound
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 13 [6 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Bowel Wall Thickness (BWT)
Description: Change in Bowel Wall Thickness at week 14 as compared to baseline, prior to initiating infliximab (IFX 0).
Time Frame: Baseline and Week 14
Measure: Median (Full Range); unit: mm
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
mm
  baseline | 5 [1 to 7]
  week 14 | 4 [2 to 7]

2. Primary Outcome: Change in Weighted Pediatric Crohn's Disease Activity Index (wPCDAI)
Description: wPCDAI at week 14 as compared to baseline. PCDAI includes three history items (abdominal pain, number of liquid stools, general wellbeing), five physical examination items (abdominal examination, perirectal disease, extraintestinal manifestations, weight, height), and three laboratory tests (hematocrit, albumin, erythrocyte sedimentation rate). Items are scored on a three-point scale (zero, 5, or 10 points) except for hematocrit and erythrocyte sedimentation rate which are scored as zero, 2.5 or 5 points. PCDAI scores can range from zero to 125 with higher scores indicating more active disease.
Time Frame: Baseline and Week 14
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
score on a scale
  baseline | 17.5 [7.5 to 85]
  week 14 | 0 [0 to 10]

3. Secondary Outcome: Change in Fecal Calprotectin
Description: change in fecal calprotectin at week 14 compared to baseline, using a specimen collection kit given to subjects
Time Frame: Baseline and Week 14
Measure: Median (Full Range); unit: mcg/g
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
mcg/g
  baseline | 358 [16 to 1074]
  week 14 | 246 [16 to 974]

4. Secondary Outcome: C-Reactive Protein
Description: C-Reactive Protein (CRP) blood level
Time Frame: 14 weeks
Measure: Median (Full Range); unit: mg/L
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
mg/L
  baseline | 16.7 [0.6 to 121]
  week 14 | 2.5 [0.2 to 23]

5. Secondary Outcome: Change in Erythrocyte Sedimentation Rate (ESR)
Description: Change in Erythrocyte Sedimentation Rate (ESR) blood level at Week 14 from baseline
Time Frame: baseline and 14 weeks
Measure: Median (Full Range); unit: mm/hr
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
mm/hr
  baseline | 30 [3 to 81]
  week 14 | 10 [5 to 32]

6. Secondary Outcome: IFX Level
Description: Infliximab drug (IFX) level at week 14. normal levels are <0.4 µg/mL
Time Frame: Week 14
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
µg/mL | 10.8 [2.3 to 20.5]

7. Secondary Outcome: Anti-infliximab Antibodies (ATI)
Description: Anti-infliximab antibodies at week 14.
Time Frame: Week 14
Measure: Median (Full Range); unit: U/mL
Arm/Group | Small Bowel Ultrasound
Number analyzed (Participants) | 13
U/mL | 0 [0 to 8.3]

ADVERSE EVENTS:
Time Frame: 16 months
Description: based on ICH and EU Guidelines on Pharmacovigilance for Medicinal Products for Human Use
Arm/Group | Small Bowel Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Principal Investigator and the Sponsor (and its agents) that allows study results to be posted to clinicaltrials.gov, and has limitations regarding PI's rights to publications and presentations.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02488005/Prot_SAP_000.pdf